CLINICAL TRIAL: NCT04328974
Title: The Effect of Lumbar Cerebrospinal Fluid Drainage on the Neurologic Outcome Improvement in Out of Hospital Cardiac Arrest Patients Underwent Targeted Temperature Management
Brief Title: The Effect of Lumbar CSF Drainage on the Neurologic Outcome Improvement in OHCA Underwent TTM
Status: Completed | Type: Observational
Sponsor: Chungnam National University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Sponsor
Other Study IDs: 201907033003
Record Dates: First submitted 2020-03-24; First posted 2020-04-01 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-09

CONDITIONS: Heart Arrest, Out-Of-Hospital; Brain Swelling
Keywords: lumbar; intracranial pressure
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Brain Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- the lumbar CSF drainage group: We named the patients treated with the protocol and the lumbar CSF drainage as the lumbar CSF drainage group.
  Interventions: Procedure: lumbar CSF drainage

INTERVENTIONS:
Procedure: lumbar CSF drainage — We have performed the lumbar CSF drainage on the level of the lumbar spine between L3 and L4 with the patient lying in the lateral decubitus position with hips and knees flexed. A lumbar drainage catheter was inserted using a HermeticTM lumbar accessory kit (Integra Neurosciences, Plainsboro, NJ, USA) in the patients. ICP monitoring via lumbar drainage catheter was practiced using the LiquoGuard® (Möller Medical GmbH & Co KG, Fulda, Germany). ICP control strategies was initiated when ICP exceeded 15 mmHg in the absence of noxious stimuli at the rate of 10~20 ml/h via a lumbar drainage catheter until ICP was less than 15 mmHg [14, 15].

SUMMARY:
Aim: The investigators aim to evaluate the effect of lumbar cerebrospinal fluid (CSF) drainage on neurologic outcome in post-cardiac arrest (CA) patients treated with target temperature management (TTM).

Methods: This is a prospective single-center study conducted from May 2020 to November 2021 on patients who have been treated with TTM following CA. The propensity score matching is proceeded between the lumbar CSF drainage and non-lumbar CSF drainage groups. The good outcome group is defined as a Glasgow-Pittsburgh cerebral performance categories (CPC) scale 1 or 2, and the poor outcome group as a CPC between 3 and 5. Lumbar CSF drainage is initiated when intracranial pressure (ICP) exceeded 15 mmHg in the absence of noxious stimuli at the rate of 10~20 ml/h via a lumbar drainage catheter until ICP is less than 15 mmHg. The magnetic resonance imaging (MRI) is obtained between 72-96 h after return of spontaneous circulation (ROSC) to evaluate the effect of lumbar CSF drainage on attenuation of brain swelling through quantitative analysis of apparent diffusion coefficient (ADC). Multivariate logistic regression and Kaplan-Meier models are built to identify the effect of CSF drainage on the neurologic outcome improvement.

DETAILED DESCRIPTION:
1. Introduction: Global cerebral ischaemic-reperfusion brain injury following cardiac arrest (CA) can lead to intracranial hypertension and, occasionally, acute brain swelling. Even small increases in brain volume due to edema can result in harmful increases in intracranial pressure due to the brain's rigid encasement. The previous studies demonstrated a higher intracranial pressure (ICP) was strongly associated with and seemed predictive of a poor outcome, and higher ICP following global cerebral ischaemia immediately after return of spontaneous circulation (ROSC), and severe blood-brain barrier (BBB) disruption began at 24 h after ROSC in the poor neurologic outcome group treated with target temperature management (TTM).

   Several therapeutic approaches have been established for the treatment of increased ICP in traumatic brain injury, including TTM, elevation of the head, sedation, volume resuscitation, maintenance of adequate arterial oxygenation, cerebrospinal fluid drainage via a ventriculostomy, moderate hyperventilation, and mannitol administration. However, despite these various therapies, a considerable number of patients remain nonresponsive to aggressive management strategies. During the last decades, controlled lumbar cerebrospinal fluid (CSF) drainage has been considered to be contraindicated in the setting of increased ICP because of the possibility of transtentorial or tonsillar herniation. In contrast, a recent report on the use of lumbar CSF drainage to treat refractory increased ICP suggested that this controversial therapeutic strategy might be efficient and a valuable treatment when applied to carefully selected patients had discernible basal cisterns and controlled release of CSF under monitoring of ICP and vital signs. Plus, much of the CSF volume is present in the subarachnoid spaces and cisterns around the brain. This CSF is not accessible for drainage by ventriculostomies but is accessible by lumbar drainage.

   However, to the best of our knowledge, there is no study on the effect of lumbar CSF drainage to improve neurologic outcome in CA patients treated with TTM. The investigators aim to evaluate the effect of lumbar CSF drainage on neurologic outcome in post-CA patients treated with TTM.
2. Methods: This study was approved by the Institutional Review Board of the Chungnam National University Medical Centre (CNUH IRB 2019-07-033-003). The investigators will obtain approval and consent from the next of kin before enrolment.

2.1. Study design and patients: This is a prospective single-center study conducted from May 2020 to November 2021 on patients who have been treated with TTM following OHCA. The primary endpoint is to measure the effect of the lumbar CSF drainage on the neurologic outcome using the Glasgow-Pittsburgh cerebral performance categories (CPC) scale in post-CA patients treated with TTM. The secondary endpoint is to measure the effect of the lumbar CSF drainage on attenuation of brain edema using MRI in post-CA patients treated with TTM. The data are collected from the electrical medical record. The investigators name the patients are treated with our standard protocol as the non-lumbar CSF drainage group, whereas the patients treated with the protocol and the lumbar CSF drainage are called as the lumbar CSF drainage group. The investigators measure neurological out-comes 6 months after ROSC using CPC scale, either through face-to-face interviews or structured telephone interviews. Phone interviews will be undertaken by an emergency physician who is fully informed of the protocol and blinded to the patient's prognosis. The CPC score classifies patients into 5 categories: CPC 1 (good performance), CPC 2 (moderate disability), CPC 3 (severe disability), CPC 4 (vegetative state), or CPC 5 (brain death or death). The good outcome group is defined as a CPC 1 or 2, and the poor outcome group as a CPC between 3 and 5. Resuscitated cardiac arrest patients whose GCS is 8 or less after ROSC, and who undergo TTM are included in the study. The exclusion criteria for this study are as follows: (1) < 18 y of age, (2) traumatic CA or interrupted TTM (due to haemodynamic instability), (3) not eligible for TTM (i.e., intracranial haemorrhage, active bleeding, known terminal illness, or poor pre-arrest neurological status), (4) ineligible for LP (i.e., brain computed tomography showed severe cerebral oedema, obliteration of the basal cisterns, occult intracranial mass lesion, antiplatelet therapy, anticoagulation therapy, or coagulopathy: platelet count < 40 x 103/mL or international normalized ratio (INR) > 1.5) (5) on extracorporeal membrane oxygenation, (6) there are no next of kin to consent to LP, and (7) refusal of further treatment by the next of kin.

2.2. TTM protocol: TTM is applied using cooling devices (Arctic Sun ® Energy Transfer Pads TM, Medivance Corp., Louisville, USA). The target temperature of 33°C is maintained for 24 h with subsequent rewarming to 37°C at a rate of 0.25°C /h. Temperature is monitored using an esophageal and bladder temperature probe. ADMS™ (Anaesthetic Depth Monitor for Sedation, Unimedics CO., LTD., Seoul, Korea) is used to monitor the anaesthesia depth. Midazolam (0.05 mg/kg intravenous bolus, followed by a titrated intravenous continuous infusion at a dose between 0.05 and 0.2 mg/kg/h) and cisatracurium (0.15 mg/kg intravenous bolus, followed with an infusion of up to 0.3 mg/kg/h) are administered for sedation and control of shivering. Electroencephalography is performed if there is a persistent deterioration of the patient's level of consciousness, involuntary movements, or seizures. If there is evidence of electrographic seizure or a clinical diagnosis of seizure, anti-epileptic drugs are administered; levetiracetam (loading dose 2 g bolus intravenously and maintenance dose, 1 g bolus twice daily, intravenously). Fluid resuscitation or vasopressors are administered when necessary to maintain mean arterial pressure between 85- and 100-mm Hg.

2.3. Data collection: The following data are collected from the database: age, sex, presence of a witness at the time of the collapse, bystander cardiopulmonary resuscitation (CPR), first monitored rhythm, etiology of cardiac arrest, time from collapse to CPR (no flow time), time from CPR to ROSC (low flow time), sequential organ failure assessment (SOF) score, ICP measured on immediate after ROSC, time from ROSC to inserting a lumbar drainage catheter placed through the lumbar vertebral interspace into the subarachnoid space (ICP time), and CPC at 6 months after ROSC.

2.4. ICP control via lumbar CSF drainage: The investigators have performed the lumbar CSF drainage on the level of the lumbar spine between L3 and L4 with the patient lying in the lateral decubitus position with hips and knees flexed. A lumbar drainage catheter is inserted using a HermeticTM lumbar accessory kit (Integra Neurosciences, Plainsboro, NJ, USA) in the patients. ICP monitoring via lumbar drainage catheter is practiced using the LiquoGuard® (Möller Medical GmbH & Co KG, Fulda, Germany). ICP control strategies is initiated when ICP exceed 15 mmHg in the absence of noxious stimuli at the rate of 10~20 ml/h via a lumbar drainage catheter until ICP is less than 15 mmHg.

2.5. MRI protocol and analysis: The investigators have a standardised magnetic resonance imaging (MRI) protocol for non-traumatic OHCAs. MRI imaging includes diffusion weighted image (DWI), and apparent diffusion coefficient (ADC) map. The MRI is obtained between 72-96 h after ROSC. Forty contiguous DWI sections per patient are acquired using a 3T scanner (Achieva 3 T; Philips Medical System, The Netherlands). The standard of b=1000 s/mm2 is used for all DWIs. ADC maps are created from the mono-exponential calculation of DWI with a commercial software and workstation system (Leonardo MR Workplace; Siemens Medical Solutions, Erlangen, Germany). For quantitative analysis of ADC, images are processed and analysed using software (FMRIB Software Library, Release 5.0 (c) 2012, The University of Oxford) that can extract brain tissue by eliminating cranium, optic structure, and extra-cranial soft tissues. Images are retrieved in Digital Imaging and Communications in Medicine format from picture archiving and communication system servers at the hospital and are converted to NITFI format using MRIcron (http://www.nitrc.org/projects/mricron). ADC thresholds range from 0 to 2200 X 10-6 mm2/s to exclude artefacts or pure CSF. The percentage of voxels (PV) meant voxel number of brain edema is divided by total voxel number.

The % voxels of ADC values (PV):

PV of cytotoxic edema = (Voxel numbers of ADC value ( from 0 to 600 X 10-6 mm2/s))/(Voxel numbers of ADC value (from 0 to 2200 X 10-6 mm2/s))

PV of vasogenic edema = (Voxel numbers of ADC value ( from 1050 to 2200 X 10-6 mm2/s))/(Voxel numbers of ADC value (from 0 to 2200 X 10-6 mm2/s))

2.6. Statistical analysis: The investigators report continuous variables as median with interquartile range or as mean and standard deviation depending on the normal distribution. Categorical variables are reported as frequencies and percentages. The investigators perform the propensity score matching with age, sex, presence of a witness at the time of the collapse, bystander CPR, first monitored rhythm, causes of CA, no flow time, low flow time, sequential organ failure assessment (SOFA) score, and ICP on immediate after ROSC between both groups. Comparisons between the two groups are made using the chi-square test, Fisher's exact test, the Mann-Whitney U test, or two-tailed t-test. Multivariate logistic regression models are built to identify the effect of the lumbar CSF drainage on the neurologic outcome. Kaplan-Meier analysis is performed to evaluate the effect of the lumbar CSF drainage on the neurologic outcome at 6 months after ROSC. The estimated odds ratio is considered to assess risk. All statistical analyses are performed using the PASW/SPSSTM software, version 18 (IBM Inc., Chicago, USA). Results are considered significant at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Resuscitated out of hospital cardiac arrest (OHCA) patients
* OHCA patients whose GCS is 8 or less after ROSC
* OHCA patients who undergo TTM

Exclusion Criteria:

* < 18 y of age
* Traumatic CA
* Interrupted TTM due to hemodynamic instability
* Intracranial hemorrhage
* Active bleeding
* Known terminal illness
* Poor pre-arrest neurological status
* Brain computed tomography showed severe cerebral edema
* Brain computed tomography showed obliteration of the basal cisterns
* Brain computed tomography showed occult intracranial mass lesion
* Antiplatelet therapy
* Anticoagulation therapy
* Platelet count < 40,000/mL
* International normalized ratio (INR) > 1.5
* OHCA patients on extracorporeal membrane oxygenation
* There are no next of kin to consent to LP
* Refusal of further treatment by the next of kin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A previous study reported ICP on 24 h after ROSC was 189.00 ± 46.02 mmH2O in good outcome and 265.56 ± 72.43 mmH2O in poor outcome, 40 patients were needed to achieve the power of 0.90 at a significance level of 0.01 (two-sided test).
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2023-04-02 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
the effect of the lumbar CSF drainage on the neurologic outcome | 6 months after ROSC
  The primary endpoint is to mearsure the effect of the lumbar CSF drainage on the neurologic outcome using the Glasgow Pittsburgh cerebral performance category (CPC) scale in post-CA patients treated with TTM.

SECONDARY OUTCOMES:
the effect of the lumbar CSF drainage on attenuation of brain swelling | 72-96 hours after ROSC
  The secondary endpoint is to measure the effect of the lumbar CSF drainage on attenuation of brain edema using MRI in post-CA patients treated with TTM.

CONTACTS AND LOCATIONS:
Overall Officials: Yeonho You, professor, Study Director — Chungnam National University Hospital
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iida K, Satoh H, Arita K, Nakahara T, Kurisu K, Ohtani M. Delayed hyperemia causing intracranial hypertension after cardiopulmonary resuscitation. Crit Care Med. 1997 Jun;25(6):971-6. doi: 10.1097/00003246-199706000-00013. PMID 9201049
- [Background] Polderman KH. Mechanisms of action, physiological effects, and complications of hypothermia. Crit Care Med. 2009 Jul;37(7 Suppl):S186-202. doi: 10.1097/CCM.0b013e3181aa5241. PMID 19535947
- [Background] You Y, Park J, Min J, Yoo I, Jeong W, Cho Y, Ryu S, Lee J, Kim S, Cho S, Oh S, Lee J, Ahn H, Lee B, Lee D, Na K, In Y, Kwack C, Lee J. Relationship between time related serum albumin concentration, optic nerve sheath diameter, cerebrospinal fluid pressure, and neurological prognosis in cardiac arrest survivors. Resuscitation. 2018 Oct;131:42-47. doi: 10.1016/j.resuscitation.2018.08.003. Epub 2018 Aug 4. PMID 30086374
- [Background] Park JS, You Y, Min JH, Yoo I, Jeong W, Cho Y, Ryu S, Lee J, Kim SW, Cho SU, Oh SK, Ahn HJ, Lee J, Lee IH. Study on the timing of severe blood-brain barrier disruption using cerebrospinal fluid-serum albumin quotient in post cardiac arrest patients treated with targeted temperature management. Resuscitation. 2019 Feb;135:118-123. doi: 10.1016/j.resuscitation.2018.10.026. Epub 2018 Oct 26. PMID 30612965
- [Background] Carney N, Totten AM, O'Reilly C, Ullman JS, Hawryluk GW, Bell MJ, Bratton SL, Chesnut R, Harris OA, Kissoon N, Rubiano AM, Shutter L, Tasker RC, Vavilala MS, Wilberger J, Wright DW, Ghajar J. Guidelines for the Management of Severe Traumatic Brain Injury, Fourth Edition. Neurosurgery. 2017 Jan 1;80(1):6-15. doi: 10.1227/NEU.0000000000001432. PMID 27654000
- [Background] Cushing H. Some aspects of the pathological physiology of intracranial tumors. Boston Med Surg J 1909; 141:71-80.
- [Background] Nash CS. Cerebellar herniation as a cause of death. Ann Otol Rhinol Laryngol 1937; 46: 673-80.
- [Background] VERBRUGGHEN A. Spinal puncture. Surg Clin North Am. 1946 Feb:78-90. No abstract available. PMID 21015502
- [Background] Munch EC, Bauhuf C, Horn P, Roth HR, Schmiedek P, Vajkoczy P. Therapy of malignant intracranial hypertension by controlled lumbar cerebrospinal fluid drainage. Crit Care Med. 2001 May;29(5):976-81. doi: 10.1097/00003246-200105000-00016. PMID 11378607
- [Background] Manet R, Payen JF, Guerin R, Martinez O, Hautefeuille S, Francony G, Gergele L. Using external lumbar CSF drainage to treat communicating external hydrocephalus in adult patients after acute traumatic or non-traumatic brain injury. Acta Neurochir (Wien). 2017 Oct;159(10):2003-2009. doi: 10.1007/s00701-017-3290-1. Epub 2017 Aug 8. PMID 28791479
- [Background] Murad A, Ghostine S, Colohan AR. A case for further investigating the use of controlled lumbar cerebrospinal fluid drainage for the control of intracranial pressure. World Neurosurg. 2012 Jan;77(1):160-5. doi: 10.1016/j.wneu.2011.06.018. Epub 2011 Nov 15. PMID 22154151
- [Background] Engelborghs S, Niemantsverdriet E, Struyfs H, Blennow K, Brouns R, Comabella M, Dujmovic I, van der Flier W, Frolich L, Galimberti D, Gnanapavan S, Hemmer B, Hoff E, Hort J, Iacobaeus E, Ingelsson M, Jan de Jong F, Jonsson M, Khalil M, Kuhle J, Lleo A, de Mendonca A, Molinuevo JL, Nagels G, Paquet C, Parnetti L, Roks G, Rosa-Neto P, Scheltens P, Skarsgard C, Stomrud E, Tumani H, Visser PJ, Wallin A, Winblad B, Zetterberg H, Duits F, Teunissen CE. Consensus guidelines for lumbar puncture in patients with neurological diseases. Alzheimers Dement (Amst). 2017 May 18;8:111-126. doi: 10.1016/j.dadm.2017.04.007. eCollection 2017. PMID 28603768
- [Background] Song G, You Y, Jeong W, Lee J, Cho Y, Lee S, Ryu S, Lee J, Kim S, Yoo I. Vasopressor requirement during targeted temperature management for out-of-hospital cardiac arrest caused by acute myocardial infarction without cardiogenic shock. Clin Exp Emerg Med. 2016 Mar 31;3(1):20-26. doi: 10.15441/ceem.15.090. eCollection 2016 Mar. PMID 27752611
- [Background] Naito H, Isotani E, Callaway CW, Hagioka S, Morimoto N. Intracranial Pressure Increases During Rewarming Period After Mild Therapeutic Hypothermia in Postcardiac Arrest Patients. Ther Hypothermia Temp Manag. 2016 Dec;6(4):189-193. doi: 10.1089/ther.2016.0009. Epub 2016 May 23. PMID 27213805
- [Background] Sekhon MS, Griesdale DE, Ainslie PN, Gooderham P, Foster D, Czosnyka M, Robba C, Cardim D. Intracranial pressure and compliance in hypoxic ischemic brain injury patients after cardiac arrest. Resuscitation. 2019 Aug;141:96-103. doi: 10.1016/j.resuscitation.2019.05.036. Epub 2019 Jun 8. PMID 31185256
- [Background] Park JS, Cho Y, You Y, Min JH, Jeong W, Ahn HJ, Kang C, Yoo I, Ryu S, Lee J, Kim SW, Cho SU, Oh SK, Lee J, Lee IH. Optimal timing to measure optic nerve sheath diameter as a prognostic predictor in post-cardiac arrest patients treated with targeted temperature management. Resuscitation. 2019 Oct;143:173-179. doi: 10.1016/j.resuscitation.2019.07.004. Epub 2019 Jul 12. PMID 31306717
- [Background] Longstreth WT Jr, Nichol G, Van Ottingham L, Hallstrom AP. Two simple questions to assess neurologic outcomes at 3 months after out-of-hospital cardiac arrest: experience from the public access defibrillation trial. Resuscitation. 2010 May;81(5):530-3. doi: 10.1016/j.resuscitation.2010.01.011. Epub 2010 Feb 20. PMID 20172643
- [Background] Ameloot K, De Deyne C, Ferdinande B, Dupont M, Palmers PJ, Petit T, Eertmans W, Moonen C, Belmans A, Lemmens R, Dens J, Janssens S. Mean arterial pressure of 65 mm Hg versus 85-100 mm Hg in comatose survivors after cardiac arrest: Rationale and study design of the Neuroprotect post-cardiac arrest trial. Am Heart J. 2017 Sep;191:91-98. doi: 10.1016/j.ahj.2017.06.010. Epub 2017 Jun 23. PMID 28888275

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT04328974/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT04328974/ICF_001.pdf